CLINICAL TRIAL: NCT05976750
Title: Air Optix® Night and Day® Aqua Daily Wear
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CLD265-N002
Record Dates: First submitted 2023-07-26; First posted 2023-08-04 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Refractive Errors; Myopia; Hyperopia
MeSH Terms: conditions — Refractive Errors; Myopia; Hyperopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- AONDA contact lenses: Lotrafilcon A contact lenses worn daily and removed at night for cleaning and disinfection as instructed by the eye care professional
  Interventions: Device: Lotrafilcon A contact lenses
- PV2 contact lenses: Balafilcon A contact lenses worn daily and removed at night for cleaning and disinfection as instructed by the eye care professional
  Interventions: Device: Balafilcon A contact lenses

INTERVENTIONS:
Device: Lotrafilcon A contact lenses — CE-marked silicone hydrogel contact lenses for daily wear use
  Other Names: AONDA; Air Optix® Night and Day® Aqua
  Groups: AONDA contact lenses
Device: Balafilcon A contact lenses — CE-marked silicone hydrogel contact lenses for daily wear use
  Other Names: PV2; PureVision® 2
  Groups: PV2 contact lenses

SUMMARY:
The purpose of this Post-Market Clinical Follow-Up (PMCF) study is to assess long term performance and safety of Air Optix® Night and Day® Aqua (AONDA) contact lenses in a real-world setting when worn as daily wear for vision correction.

DETAILED DESCRIPTION:
This is a non-interventional/observational study designed as a retrospective chart review. Study sites will review charts within their existing database to identify subjects who wore AONDA contact lenses or PureVision® 2 (PV2) contact lenses in both eyes for approximately 1 year following their contact lens examination. The data collection period consists of any approximately 1-year timeframe since and including 2009.

The anticipated duration of the study is approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Normal eyes, as determined by the Investigator
* At the time of the 1-year visit, subject was prescribed and wearing AONDA contact lenses or PV2 contact lenses in both eyes in a daily wear modality for at least approximately 1 year without changing wear modality
* Baseline and 1-year visit charts available
* Other protocol-specified inclusion criteria may apply

Exclusion Criteria

* Any recurrent history or active anterior segment infection, inflammation, abnormality, or disease contraindicating regular contact lens wear present at Baseline
* Use of systemic or ocular medications contraindicating regular contact lens wear at Baseline
* History of refractive surgery or irregular cornea
* Other protocol-specified exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will enroll charts following a pre-identified process.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Distance visual acuity by eye | Year 1
  The subject's chart will be reviewed for distance visual acuity.
Incidence of corneal infiltrative events | Up to Year 1
  The subject's chart will be reviewed for incidences of corneal infiltrative events occurring after the baseline exam.
Incidence of microbial keratitis | Up to Year 1
  The subject's chart will be reviewed for incidences of microbial keratitis occurring after the baseline exam.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, CRD Vision Care, Study Director — Alcon Research, LLC
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No